CLINICAL TRIAL: NCT04196569
Title: Spectacle Independence After Implantation of Trifocal and Trifocal Toric Intraocular Lenses Using Intraoperative Aberrometry: A Prospective Analysis
Brief Title: Trifocal Intraocular Lens (IOL) Aberrometry Outcomes
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Sponsor
Other Study IDs: 19-05020251
Record Dates: First submitted 2019-12-10; First posted 2019-12-12 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Cataract
Keywords: trifocal lens; trifocal intraocular lens; aberrometry
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- trifocal intraocular lens
  Interventions: Device: Alcon Trifocal and Trifocal Toric Intraocular Lenses

INTERVENTIONS:
Device: Alcon Trifocal and Trifocal Toric Intraocular Lenses — Panoptix Model #TFAT00 for the UV Absorbing Trifocal IOL. Torics:
  TFAT30, TFAT40, TFAT50, TFAT60

SUMMARY:
The goal of this study is to evaluate subject outcomes and spectacle independence with intraoperative aberrometry and trifocal IOL implantation.

ELIGIBILITY:
Inclusion Criteria:

* Able to consent to study and cataract surgery
* Visually significant cataract
* Potential post-operative visual acuity of 20/25 or better
* Age 18 years or older

Exclusion Criteria:

* Ocular pathology contraindicated for trifocal IOLs including but not limited to diabetic retinopathy, age-related macular degeneration or other macular pathology, cornea guttata, corneal scarring, corneal ectasia, glaucoma with visual field loss
* Irregular astigmatism
* Prior corneal refractive surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with a diagnosis of visually-significant cataracts who meet the inclusion and exclusion criteria will be eligible for participation in this study.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2019-12-12 (Actual); Primary Completion 2022-09-13 (Actual); Study Completion 2022-09-13 (Actual)

PRIMARY OUTCOMES:
Percentage of spectacle independence (overall) | 1 month post-cataract surgery
  This will be assessed by a Visual Quality Questionnaire, an 18 question multiple choice questionnaire to assess vision-related functioning. Grading scale: 0, no difficulty; 1, a little difficulty; 2, moderate difficulty; 3, quite difficult; 4, impossible to perform. Mean value(s) will be analyzed.
Percentage spectacle independence (overall) | 3 months post-cataract surgery
  This will be assessed by a Visual Quality Questionnaire, an 18 question multiple choice questionnaire to assess vision-related functioning. Grading scale: 0, no difficulty; 1, a little difficulty; 2, moderate difficulty; 3, quite difficult; 4, impossible to perform. Mean value(s) will be analyzed.

SECONDARY OUTCOMES:
Spectacle independence for distance, intermediate and near | 1 month post-cataract surgery
  This will be assessed by a Visual Quality Questionnaire, an 18 question multiple choice questionnaire to assess vision-related functioning. Grading scale: 0, no difficulty; 1, a little difficulty; 2, moderate difficulty; 3, quite difficult; 4, impossible to perform. Mean value(s) will be analyzed.
Spectacle independence for distance, intermediate and near | 3 months post-cataract surgery
  This will be assessed by a Visual Quality Questionnaire, an 18 question multiple choice questionnaire to assess vision-related functioning. Grading scale: 0, no difficulty; 1, a little difficulty; 2, moderate difficulty; 3, quite difficult; 4, impossible to perform. Mean value(s) will be analyzed.
Spectacle independence subgroup analysis for subjects within 0.50 D spherical equivalent (SE) | 1 month post-cataract surgery
  This will be assessed by a Visual Quality Questionnaire, an 18 question multiple choice questionnaire to assess vision-related functioning. Grading scale: 0, no difficulty; 1, a little difficulty; 2, moderate difficulty; 3, quite difficult; 4, impossible to perform. Mean value(s) will be analyzed.
Spectacle independence subgroup analysis for subjects within 0.50 D spherical equivalent (SE) | 3 months post-cataract surgery
  This will be assessed by a Visual Quality Questionnaire, an 18 question multiple choice questionnaire to assess vision-related functioning. Grading scale: 0, no difficulty; 1, a little difficulty; 2, moderate difficulty; 3, quite difficult; 4, impossible to perform. Mean value(s) will be analyzed.
Binocular, uncorrected distance visual acuity for patients within 0.50 D of intended target | 3 months post-cataract surgery
  This will be measured by visual acuity
Subject satisfaction | 3 months post-cataract surgery
  This will be assessed by a Visual Quality Questionnaire, an 18 question multiple choice questionnaire to assess vision-related functioning. Grading scale: 0, no difficulty; 1, a little difficulty; 2, moderate difficulty; 3, quite difficult; 4, impossible to perform. Mean value(s) will be analyzed.
Uncorrected binocular and monocular visual acuity at all distances | 3 months post-cataract surgery
  This will be measured by visual acuity
Distribution of residual refractive error | 3 months post-cataract surgery
  This will be measured by refractive error
Contrast sensitivity (binocular) | 1 month post-cataract surgery
  This will be measured by contrast sensitivity testing
Contrast sensitivity (binocular) | 3 months post-cataract surgery
  This will be measured by contrast sensitivity testing
Percentage of subjects with <=0.50 D of refractive cylinder | 1 month post-cataract surgery
  This will be measured by refractive error
Percentage of subjects with <=0.50 D of refractive cylinder | 3 months post-cataract surgery
  This will be measured by refractive error

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Brissette, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No